CLINICAL TRIAL: NCT04102449
Title: Validation of the PsASon ULtrasound Scores in Patients With Psoriatic Arthritis Undergoing TReatment With Apremilast
Acronym: PSA-ULTRA
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Funding stopped
Sponsor: Medical University of Graz (Other)
Collaborators: Celgene Corporation (Industry); Medical University of Vienna (Other); Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AP-CL-PSA-PI-12856
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Psoriatic Arthritis
Keywords: Ultrasound; Psoriatic arthritis; Outcome measures; Apremilast; Disease activity
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — apremilast

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with Apremilast (Other): Single group:
  Apremilast will be prescribed according to the patient information leaflet, i.e.:
  Dosage form: Oral pill Dosage and Frequency: First 6 days titration phase, followed by 30mg twice daily (in case of kidney problems 30mg once daily in the morning). Treatment duration at the discretion of the treating physician.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Single arm receiving Apremilast and ultrasound examinations

SUMMARY:
The main purpose of this study is to validate the ultrasound scores PsASon22 and PsASon13 in patients with active psoriatic arthritis undergoing a treatment with Apremilast.

DETAILED DESCRIPTION:
This is a prospective, multicentre, phase IV trial assessing the value of the ultrasound scores PsASon22 and PsASon13 in differentiating between clinically active and inactive patients with psoriatic arthritis, following a treatment with Apremilast for up to 24 months. Additionally, convergent construct validity, inter/intra-reader reliability, sensitivity to change and differences in change in certain patients will be tested for the ultrasound scores.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years and <90 years of age
2. PsA according to CASPAR criteria
3. Peripheral manifestation (arthritis, tenosynovitis, dactylitis and/or enthesitis)
4. Active disease as defined by a DAPSA >14 and clinical indication for treatment with Apremilast (as per approved indication for PsA, including failure to methotrexate)
5. Written informed consent

Exclusion Criteria:

1. Inability to perform US at any site included in the PsASon22 or PsASon13 score (f.e. due to complete destruction of a joint)
2. Planned surgery within the study period or history of surgery of any of the joints to be investigated clinically or by sonography.
3. Contraindication to Apremilast (as per patient information leaflet)
4. Current severe medical illness requiring hospitalization
5. Pregnancy or lactation
6. Inability of the patient to follow the treatment protocol
7. Fulfillment of the MDA Criteria or DAPSA≤14
8. Current treatment with any investigational drug
9. Current treatment with glucocorticoids at a prednisone equivalent >10mg
10. Intra-articular glucocorticoid injection in one of the joints to be investigated clinically or by sonography, or intra-muscular glucocorticoid injection within 8 weeks before baseline
11. Change, including dosage changes or discontinuation, of csDMARD treatment (with the exception of leflunomide) in the last 4 weeks before baseline
12. Change, including dosage changes or discontinuation of leflunomide treatment in the last 8 weeks before baseline. (Exception: If patients stop leflunomide and complete an 11 day treatment with cholestyramine (8g, 3 x daily), prior to the baseline visit, they may enter the study.)
13. Current bDMARD, tsDMARD treatment
14. Prior bDMARD or tsDMARD treatment without a minimal washout period before baseline (the minimal washout period is twice the half-life of the respective drug)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
The difference in the change-score of the PsASon22 | 4-12-24 months
  The main outcome is the difference in the change-score of the PsASon22 between patients achieving low disease activity or remission (DAPSA≤14) and patients not achieving this target under a treatment with Apremilast.
  The Psoratic Arthritis Sonography Score 22, PsASon22 (range 0-260), is a sum score, including grey scale and power doppler measurements of 22 joints (6 MCPs, 4-H-PIPs, 2 MTPs, 4 H-DIPs, 2 F-DIPs, 4 large joints) and 4 entheses (lateral epicondyle and distal patella - bilateral), with a higher score presumably indicating higher disease activity.
The difference in the change-score of the PsASon13 | 4-12-24 months
  The main outcome is the difference in the change-score of the PsASon13 between patients achieving low disease activity or remission (DAPSA≤14) and patients not achieving this target under a treatment with Apremilast.
  The Psoratic Arthritis Sonography Score 13, PsASon13 (range 0-134), is a sum score, including grey scale and power doppler measurements of 13 joints (2 MCPs, 3-H-PIPs, 1-F-PIP, 2 MTPs, 1 H-DIPs, 2 F-DIPs, 2 large joints) and 2 entheses (lateral epicondyle and distal patella - unilateral), with a higher score presumably indicating higher disease activity.

SECONDARY OUTCOMES:
Convergent construct validity of PsAson22 and PsASon13 | 4-12-24 months
  Convergent construct validity will be assessed by correlating the ultrasound scores to clinical composite scores (f.e. DAPSA)
Sensitivity to Change of PsASon22 and PsASon13 | 4-12-24 months
  Sensitivity to change will be assessed by measuring the PsASon22 and PsASon 13 scores at four different time points (Baseline and after 4, 12 and 24 months)
Interrater reliability of PsASon22 and PsASon13 | 4-12-24 months
  Interrater reliability will be assessed by performing multiple ultrasound examinations for one patient by multiple examinators
Intrarater reliability of PsASon22 and PsASon13 | 4-12-24 months
  Intrarater reliability will be assessed by performing multiple ultrasound examinations for one patient by multiple examinators
Differences in PsASon22 and PsASon13 change | 4-12-24 months
  Differences in change will be assessed by comparing the change scores of patients with initially high disease activity (DAPSA>28) with the change scores of patients with initially moderate disease activity (DAPSA>14-≤28)

CONTACTS AND LOCATIONS:
Overall Officials: Rusmir Husic, Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria